CLINICAL TRIAL: NCT00010335
Title: A Pilot Study of High-Dose Immunosuppression Followed by Infusion of CD34-Selected Autologous or Syngeneic Peripheral Blood Stem Cells for Treatment of Refractory Autoimmune Disorders
Brief Title: Pilot Study of Total Body Irradiation in Combination With Cyclophosphamide, Anti-thymocyte Globulin, and Autologous CD34-Selected Peripheral Blood Stem Cell Transplantation in Children With Refractory Autoimmune Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1353.00; FHCRC-1353.00; 199/15575 (Other: ORD)
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Systemic Sclerosis; Systemic Lupus Erythematosus; Dermatomyositis; Juvenile Rheumatoid Arthritis; Autoimmune Diseases
Keywords: arthritis & connective tissue diseases; dermatomyositis; immunologic disorders and infectious disorders; juvenile rheumatoid arthritis; rare disease; systemic lupus erythematosus; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Lupus Erythematosus, Systemic; Dermatomyositis; Arthritis, Juvenile; Autoimmune Diseases; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive a stem cell transplant.
  Interventions: Procedure: Stem Cell Transplantation; Device: CD34 selection

INTERVENTIONS:
Procedure: Stem Cell Transplantation — Participants will receive a stem cell transplantation along with irradiation and the drugs anti-thymocyte globulin, cyclophosphamide, and filgrastim as noted in the text of this record.
Device: CD34 selection — CD34+ cells are separated from the rest of the peripheral blood stem cells.

SUMMARY:
OBJECTIVES: I. Determine the safety and long term complications of total body irradiation in combination with cyclophosphamide, anti-thymocyte globulin, and autologous CD34-selected peripheral blood stem cell (PBSC) transplantation in children with refractory autoimmune disorders.

II. Determine the efficacy of this treatment regimen in these patients. III. Determine the reconstitution of immunity after autologous CD34-selected PBSC transplantation in these patients.

IV. Determine engraftment of autologous CD34-selected PBSC in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a multicenter study. Patients receive filgrastim (G-CSF) subcutaneously daily until peripheral blood stem cell (PBSC) collection is completed. CD34+ cells are separated from the rest of the PBSCs.

Patients undergo total body irradiation twice daily on days -5 and -4. Patients receive anti-thymocyte globulin IV on days -5, -3, -1, 1, 3, and 5 and cyclophosphamide IV on days -3 and -2. CD34-selected PBSCs are reinfused on day 0. Patients receive G-CSF IV daily beginning on day 0 and continuing until blood counts recover.

Patients are followed annually for 5 years and then every 5 years thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of 1 of the following based on American College of Rheumatology (ACR) Criteria: Severe juvenile rheumatoid arthritis (systemic onset or polyarticular course) Juvenile systemic lupus erythematosus Systemic sclerosis Dermatomyositis
* Refractory to standard or aggressive therapy OR unacceptable toxicity from standard therapy
* Reasonable expectation of possible improvement as evidenced by a good potential for rehabilitation therapy and adequate social factors
* No serious CNS damage that would preclude significant functional recovery

--Prior/Concurrent Therapy--

* Chemotherapy: At least 4 weeks since prior methotrexate or cyclophosphamide
* Endocrine therapy: At least 4 weeks since prior intra-arterial steroids Juvenile rheumatoid arthritis patients should continue steroids without taper throughout mobilization and harvest of stem cells If receiving corticosteroids, must be continued without taper

Other:

* At least 4 weeks since prior anti-inflammatory agents such as non-steroidal anti-inflammatory drugs (NSAIDs) or sulfasalazine
* At least 4 weeks since prior cyclosporine, tacrolimus, mycophenolate mofetil, azathioprine, penicillamine, or etanercept

--Patient Characteristics--

* Life expectancy: At least 30 days
* Hematopoietic: Absolute neutrophil count at least 1,000/mm3 OR Platelet count at least 100,000/mm3 No bone marrow aspirate or biopsy consistent with production defect (depletion of neutrophil precursors or megakaryocytes) No myelodysplasia
* Hepatic: Bilirubin no greater than 2.5 mg/dL AST no greater than 300 U/L on two sequential tests No severe liver dysfunction within past month No active hepatitis A, B, or C
* Renal: No end-stage glomerulonephritis or renal disease Creatinine clearance at least 40 mL/min
* Cardiovascular: No uncontrolled malignant arrhythmia No New York Heart Association class III or IV congestive heart failure Ejection fraction at least 50%
* Pulmonary: DLCO at least 45% (DLCO at least 70% for patients with pulmonary disease caused by documented processes other than primary autoimmune disorder, such as infectious pneumonia or aspiration pneumonia) No severe pulmonary hypertension (PAP greater than 50) without potential for significant improvement

Other:

* No medical or psychosocial reasons that would make hematopoietic stem cell collection intolerable
* No increased anesthetic risks
* No fever higher than 39 degrees C
* No positive serology for toxoplasmosis
* No active life threatening infection not responsive to therapy
* No other disease or organ dysfunction that would limit survival
* No known hypersensitivity to murine or equine proteins
* No known primary immunodeficiency disease HIV negative

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2000-11; Primary Completion 2010-07 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mortality | Annually for 5 years and then every 5 years thereafter

SECONDARY OUTCOMES:
Immune reconstitution, engraftment, efficacy, late-effects | Annually for 5 years and then every 5 years thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Ann Woolfrey, Study Chair — Fred Hutchinson Cancer Center; Carol A. Wallace, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States